CLINICAL TRIAL: NCT03412747
Title: A Phase 3, Multicenter, Randomized, Double-Blind Study With an Active-Controlled Initial Treatment Period Followed by a Dose-Blind Maintenance Treatment Period to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of Bimekizumab in Adult Subjects With Moderate to Severe Chronic Plaque Psoriasis
Acronym: BE SURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PS0008; 2016-003392-22 (EudraCT Number)
Record Dates: First submitted 2018-01-22; First posted 2018-01-26 (Actual); Results first posted 2022-03-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Plaque Psoriasis; Moderate to Severe Plaque Psoriasis
Keywords: Bimekizumab; PSO; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bimekizumab Arm 1 (Experimental): Subjects will receive bimekizumab dose regimen 1 for 56 weeks. Subjects will receive placebo at pre-specified time-points to maintain the blinding.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Bimekizumab Arm 2 (Experimental): Subjects will receive bimekizumab dose regimen 1 for 16 weeks and will proceed with bimekizumab dose regimen 2 until week 56. Subjects will receive placebo at pre-specified time-points to maintain the blinding.
  Interventions: Drug: Bimekizumab; Other: Placebo
- Adalimumab Arm (Active Comparator): Subjects will receive adalimumab for 24 weeks and will then receive bimekizumab dose regimen 1 until week 56. Subjects will receive placebo at pre-specified time-points to maintain the blinding.
  Interventions: Drug: Bimekizumab; Drug: Adalimumab; Other: Placebo

INTERVENTIONS:
Drug: Bimekizumab — Subjects will receive bimekizumab at pre-defined timepoints in dose regimen 1 and/or dose regimen 2.
  Other Names: UCB4940
Drug: Adalimumab — Adalimumab will be administered according to the labeling recommendations.
  Other Names: Humira®
  Arms: Adalimumab Arm
Other: Placebo — Subjects will receive Placebo at pre-specified time points to maintain the blinding of the Investigational Medicinal Products (IMP).
  Other Names: PBO

SUMMARY:
This is a study to compare the efficacy of bimekizumab versus adalimumab in the treatment of subjects with moderate to severe chronic plaque psoriasis (PSO).

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Chronic plaque PSO for at least 6 months prior to the Screening Visit
* Psoriasis Area Severity Index (PASI) >=12 and body surface area (BSA) affected by PSO >=10% and Investigator's Global Assessment (IGA) score >=3 on a 5-point scale
* Subject is a candidate for systemic PSO therapy and/or phototherapy
* Female subject of child bearing potential must be willing to use highly effective method of contraception

Exclusion Criteria:

* Subject has a known hypersensitivity to any excipients of bimekizumab or adalimumab
* Subject has an active infection (except common cold), a serious infection, or a history of opportunistic or recurrent chronic infections
* Subject has concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection
* Subject has known tuberculosis (TB) infection, is at high risk of acquiring TB infection, or has current or history of nontuberculous mycobacterium (NTMB) infection
* Subject has any other condition, including medical or psychiatric, which, in the Investigator's judgment, would make the subject unsuitable for inclusion in the study
* Subject has had previous exposure to adalimumab
* Presence of active suicidal ideation or positive suicide behavior
* Presence of moderately severe major depression or severe major depression
* Subject has any active malignancy or history of malignancy within 5 years prior to the Screening Visit EXCEPT treated and considered cured cutaneous squamous or basal cell carcinoma, or in situ cervical cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (77):
- United States (23):
  - Ps0008 957, Glendale, Arizona
  - Ps0008 927, Los Angeles, California
  - Ps0008 955, San Diego, California
  - Ps0008 943, San Luis Obispo, California
  - Ps0008 967, Santa Monica, California
  - Ps0008 939, Danbury, Connecticut
  - Ps0008 934, Washington D.C., District of Columbia
  - Ps0008 906, Boca Raton, Florida
  - Ps0008 936, Tampa, Florida
  - Ps0008 900, West Des Moines, Iowa
  - Ps0008 905, Overland Park, Kansas
  - Ps0008 940, Beverly, Massachusetts
  - Ps0008 925, Brighton, Massachusetts
  - Ps0008 917, Troy, Michigan
  - Ps0008 908, East Windsor, New Jersey
  - Ps0008 961, Rocky Mount, North Carolina
  - Ps0008 935, Winston-Salem, North Carolina
  - Ps0008 932, Oklahoma City, Oklahoma
  - Ps0008 929, Portland, Oregon
  - Ps0008 945, Greer, South Carolina
  - Ps0008 931, Dallas, Texas
  - Ps0008 924, Houston, Texas
  - Ps0008 951, Houston, Texas
- Australia (6):
  - Ps0008 008, East Melbourne
  - Ps0008 004, Fremantle
  - Ps0008 007, Hectorville
  - Ps0008 010, Kogarah
  - Ps0008 005, Phillip
  - Ps0008 009, Woolloongabba
- Canada (10):
  - Ps0008 659, Calgary
  - Ps0008 663, Mississauga
  - Ps0008 660, Montreal
  - Ps0008 661, Peterborough
  - Ps0008 662, Toronto
  - Ps0008 664, Toronto
  - Ps0008 657, Waterloo
  - Ps0008 669, Windsor
  - Ps0008 670, Windsor
  - Ps0008 674, Winnipeg
- Germany (9):
  - Ps0008 207, Berlin
  - Ps0008 218, Bonn
  - Ps0008 203, Dresden
  - Ps0008 211, Hamburg
  - Ps0008 220, Hamburg
  - Ps0008 215, Lübeck
  - Ps0008 213, Mahlow
  - Ps0008 205, Osnabrück
  - Ps0008 217, Schweinfurt
- Hungary (6):
  - Ps0008 252, Budapest
  - Ps0008 254, Budapest
  - Ps0008 255, Budapest
  - Ps0008 256, Debrecen
  - Ps0008 251, Gyula
  - Ps0008 260, Szeged
- Poland (16):
  - Ps0008 355, Bialystok
  - Ps0008 362, Bialystok
  - Ps0008 371, Bydgoszcz
  - Ps0008 352, Gdansk
  - Ps0008 359, Katowice
  - Ps0008 366, Katowice
  - Ps0008 363, Krakow
  - Ps0008 360, Lodz
  - Ps0008 372, Lodz
  - Ps0008 356, Lublin
  - Ps0008 364, Nowa Sól
  - Ps0008 353, Szczecin
  - Ps0008 354, Warsaw
  - Ps0008 365, Wroclaw
  - Ps0008 367, Wroclaw
  - Ps0008 373, Wroclaw
- Russia (3):
  - Ps0008 405, Saint Petersburg
  - Ps0008 401, Saratov
  - Ps0008 406, Yaroslavl
- South Korea (2):
  - Ps0008 702, Gwangju
  - Ps0008 700, Seoul
- Taiwan (2):
  - Ps0008 754, Taipei
  - Ps0008 755, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: http://www.Vivli.org

REFERENCES:
- [Result] Thaci D, Vender R, de Rie MA, Conrad C, Pariser DM, Strober B, Vanvoorden V, Wang M, Madden C, de Cuyper D, Kimball AB. Safety and efficacy of bimekizumab through 2 years in patients with moderate-to-severe plaque psoriasis: longer-term results from the BE SURE randomized controlled trial and the open-label extension from the BE BRIGHT trial. Br J Dermatol. 2023 Jan 23;188(1):22-31. doi: 10.1093/bjd/ljac021. PMID 36689515
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Stein Gold L, Merola JF, Peterson L, Wixted K, Cross N, Deherder D, Thaci D. Bimekizumab Safety in Patients With Moderate to Severe Plaque Psoriasis: Pooled Results From Phase 2 and Phase 3 Randomized Clinical Trials. JAMA Dermatol. 2022 Jul 1;158(7):735-744. doi: 10.1001/jamadermatol.2022.1185. PMID 35544084
- [Result] Gordon KB, Langley RG, Warren RB, Okubo Y, Rosmarin D, Lebwohl M, Peterson L, Madden C, de Cuyper D, Davies O, Thaci D. Bimekizumab safety in patients with moderate-to-severe plaque psoriasis: pooled data from up to 3 years of treatment in randomized phase III trials. Br J Dermatol. 2024 Mar 15;190(4):477-485. doi: 10.1093/bjd/ljad429. PMID 37950894
- [Result] Strober B, Boehncke WH, Krueger JG, Magnolo N, Vender R, Warren RB, Lopez Pinto JM, Kavanagh S, Hoepken B, Gisondi P. Bimekizumab Efficacy in Psoriasis by Subgroups: Post Hoc Analysis of Phase 3/3b Clinical Trials. Dermatol Ther (Heidelb). 2025 Dec;15(12):3633-3650. doi: 10.1007/s13555-025-01557-1. Epub 2025 Oct 8. PMID 41060492
- [Result] Armstrong A, Papp KA, Lebwohl M, Savage LJ, Yamanaka K, Vlase DE, Warham R, Lambert J, Lopez Pinto JM, Wixted K, Thaci D. Bimekizumab Impact on Patient-Reported Outcomes in Plaque Psoriasis: 4-Year Results from BE SURE, BE VIVID, BE READY, and BE BRIGHT. Dermatol Ther (Heidelb). 2025 Dec 8. doi: 10.1007/s13555-025-01595-9. Online ahead of print. PMID 41359217
- [Derived] Merola JF, Warren RB, Thaci D, Gordon KB, Nishida E, Strober B, Conrad C, Kavanagh S, Lopez Pinto JM, Hoepken B, Gisondi P. Bimekizumab Complete Clearance of Both Skin and Nail Psoriasis: Comparative Efficacy in Phase III/IIIb Studies. Am J Clin Dermatol. 2025 Nov;26(6):967-979. doi: 10.1007/s40257-025-00968-2. Epub 2025 Aug 31. PMID 40886218
- [Derived] Merola JF, Gottlieb AB, Pinter A, Elewski B, Gooderham M, Warren RB, Piaserico S, Wixted K, Cross N, Tilt N, Wiegratz S, Mrowietz U. Bimekizumab Efficacy in High-Impact Areas: Pooled 2-Year Analysis in Scalp, Nail, and Palmoplantar Psoriasis from Phase 3/3b Randomized Controlled Trials. Dermatol Ther (Heidelb). 2024 Dec;14(12):3291-3306. doi: 10.1007/s13555-024-01295-w. Epub 2024 Nov 22. PMID 39578348
- [Derived] Kokolakis G, Warren RB, Strober B, Blauvelt A, Puig L, Morita A, Gooderham M, Korber A, Vanvoorden V, Wang M, de Cuyper D, Madden C, Nunez Gomez N, Lebwohl M. Bimekizumab efficacy and safety in patients with moderate-to-severe plaque psoriasis who switched from adalimumab, ustekinumab or secukinumab: results from phase III/IIIb trials. Br J Dermatol. 2023 Feb 22;188(3):330-340. doi: 10.1093/bjd/ljac089. PMID 36751950
- [Derived] Warren RB, Blauvelt A, Bagel J, Papp KA, Yamauchi P, Armstrong A, Langley RG, Vanvoorden V, De Cuyper D, Cioffi C, Peterson L, Cross N, Reich K. Bimekizumab versus Adalimumab in Plaque Psoriasis. N Engl J Med. 2021 Jul 8;385(2):130-141. doi: 10.1056/NEJMoa2102388. Epub 2021 Apr 23. PMID 33891379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in January 2018 and concluded in February 2020.
Pre-assignment Details: This study included 4 periods: a Screening Period (2 to 5 weeks), an Initial Treatment Period (16 weeks), a Maintenance Treatment Period (40 weeks), and a Safety Follow-Up (SFU) Visit (20 weeks after the final dose of study drug). Participant Flow refers to the Randomized Set.
Groups:
- Bimekizumab 320 Milligrams (mg) Q4W/Q8W: Study participants received bimekizumab 320 mg Q4W for 16 weeks and proceeded with bimekizumab 320 mg Q8W until Week 56. Study participants received placebo at pre-specified time-points to maintain the blinding.
- Bimekizumab 320 mg Q4W: Study participants received bimekizumab 320 mg Q4W for 56 weeks. Study participants received placebo at pre-specified time-points to maintain the blinding.
- Adalimumab: Study participants received adalimumab for 24 weeks and then received bimekizumab 320 mg Q4W until Week 56. Study participants received placebo at pre-specified time-points to maintain the blinding.
Period: Initial Treatment Period: Wk0-Wk16
Arm/Group | Bimekizumab 320 Milligrams (mg) Q4W/Q8W | Bimekizumab 320 mg Q4W | Adalimumab
Started | 161 | 158 | 159
Completed | 154 | 153 | 150
Not Completed | 7 | 5 | 9
Not completed — Adverse Event | 2 | 2 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 2 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Participant moved out of state | 1 | 0 | 0
Period: Maintenance Treatment Period: Wk16-Wk24
Arm/Group | Bimekizumab 320 Milligrams (mg) Q4W/Q8W | Bimekizumab 320 mg Q4W | Adalimumab
Started | 154 | 153 | 150
Completed | 149 | 152 | 149
Not Completed | 5 | 1 | 1
Not completed — Adverse Event | 3 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Maintenance Treatment Period: Wk24-Wk56
Arm/Group | Bimekizumab 320 Milligrams (mg) Q4W/Q8W | Bimekizumab 320 mg Q4W | Adalimumab
Started | 149 | 152 | 149
Completed | 143 | 143 | 133
Not Completed | 6 | 9 | 16
Not completed — Adverse Event | 3 | 4 | 6
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 2 | 5
Not completed — Withdrawal by Subject | 3 | 1 | 4
Not completed — Moving out of town | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Randomized Set (RS) which consisted of all randomized study participants.
Arm/Group | Bimekizumab 320 Milligrams (mg) Q4W/Q8W | Bimekizumab 320 mg Q4W | Adalimumab | Total Title
Number analyzed (Participants) | 161 | 158 | 159 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 2 | 5
  Between 18 and 65 years | 145 | 147 | 137 | 429
  >=65 years | 13 | 11 | 20 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (13.5) | 45.3 (13.2) | 45.5 (14.3) | 44.9 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 56 | 45 | 150
  Male | 112 | 102 | 114 | 328
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 13 | 10 | 11 | 34
  Black or African American | 2 | 2 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  White | 140 | 140 | 141 | 421
  Other/Mixed | 4 | 5 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 90 (PASI90) Response at Week 16
Description: The PASI90 response assessments are based on at least 90% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of respective section, and weighted by the percentage of the person's affected skin for respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: The Randomized Set (RS) consisted of all randomized study participants. Both BKZ 320 mg Q4W and BKZ 320 mg Q4W/Q8W arms are identical in terms of treatment received until Week 16 and therefore they are combined for analyses.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS): This group consisted of participants from both bimekizumab 320 mg Q4W and bimekizumab 320 mg Q8W who received bimekizumab 320 mg Q4W for 16 weeks. Participants formed the Randomized Set (RS).
- Adalimumab (RS): Study participants received adalimumab for 24 weeks and then received bimekizumab 320 mg Q4W until Week 56. Study participants received placebo at pre-specified time-points to maintain the blinding. Participants formed the Randomized Set (RS).
Arm/Group | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 319 | 159
percentage of participants | 86.2 | 47.2
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); Risk Difference: BKZ-ADA calculated using stratified CMH; Test type: Non-Inferiority — The evaluation of non-inferiority is tested at a 1-sided alpha level of 0.025 and based on a 1-sided 97.5% CI and a non-inferiority margin of 10%; Risk Difference (RD) = 39.3, 95% CI 2-sided [30.9 to 47.7]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); Odds ratio: BKZ/ADA calculated using stratified Cochran-Mantel-Haenszel (CMH) test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 7.459, 95% CI 2-sided [4.709 to 11.816]

2. Primary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Response (Clear or Almost Clear With at Least 2-Category Improvement Relative to Baseline) at Week 16
Description: The IGA measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] or almost clear [1] with at least a two-category improvement from Baseline at Week 16.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 319 | 159
percentage of participants | 85.3 | 57.2
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); Risk Difference: BKZ-ADA calculated using stratified CMH; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Risk Difference (RD) = 28.2, 95% CI 2-sided [19.7 to 36.7]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 4.341, 95% CI 2-sided [2.785 to 6.765]

3. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 24
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 24
Population: The Randomized Set (RS) consisted of all randomized study participants. BKZ 320 mg Q4W and BKZ 320 mg Q4W/Q8W arms were also combined for analyses purposes at Week 24 since they differ only one dose (Week 20).
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 320 mg Q4W/Q8W (RS): Study participants received bimekizumab 320 mg Q4W for 16 weeks and proceeded with bimekizumab 320 mg Q8W until Week 56. Study participants received placebo at prespecified time-points to maintain the blinding. Participants formed the Randomized Set (RS).
- Bimekizumab 320 mg Q4W (RS): Study participants received bimekizumab 320 mg Q4W for 56 weeks. Study participants received placebo at pre-specified time-points to maintain the blinding. Participants formed the Randomized Set (RS).
Arm/Group | Bimekizumab 320 mg Q4W/Q8W (RS) | Bimekizumab 320 mg Q4W (RS) | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 161 | 158 | 319 | 159
percentage of participants | 85.1 | 86.1 | 85.6 | 51.6
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 6.231, 95% CI 2-sided [3.515 to 11.046]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); Odds ratio: BKZ/ADA calculated using stratified CMH test with region and prior biologic exposure as stratification variables; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 5.750, 95% CI 2-sided [3.657 to 9.041]

4. Secondary Outcome: Percentage of Participants With an IGA Response (Clear or Almost Clear With at Least 2-category Improvement Relative to Baseline) at Week 24
Description: The IGA measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0= clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1= almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2= mild thickening, pink to light red coloration and predominately fine scaling, 3= moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4= severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0] with at least a two-category improvement from Baseline at Week 24.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W/Q8W (RS) | Bimekizumab 320 mg Q4W (RS) | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 161 | 158 | 319 | 159
percentage of participants | 87.0 | 86.1 | 86.5 | 57.9
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 4.724, 95% CI 2-sided [2.683 to 8.318]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 4.762, 95% CI 2-sided [3.014 to 7.523]

5. Secondary Outcome: Percentage of Participants With a PASI75 Response at Week 4
Description: The PASI75 response assessments are based on at least 75% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 4
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 319 | 159
percentage of participants | 76.5 | 31.4
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 7.103, 95% CI 2-sided [4.637 to 10.880]

6. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 16
Description: The PASI100 response assessments are based on a 100% improvement in PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 319 | 159
percentage of participants | 60.8 | 23.9
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 4.974, 95% CI 2-sided [3.230 to 7.661]

7. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 24
Description: The PASI100 response assessments are based on a 100% improvement in the PASI score from Baseline. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. The minimum possible PASI score is 0= no disease, the maximum score is 72= maximal disease.
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W/Q8W (RS) | Bimekizumab 320 mg Q4W (RS) | Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) | Adalimumab (RS)
Number analyzed (Participants) | 161 | 158 | 319 | 159
percentage of participants | 65.8 | 67.7 | 66.8 | 29.6
Statistical Analysis 1: Comparison: Bimekizumab 320 mg Q4W (RS) vs Adalimumab (RS); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 5.249, 95% CI 2-sided [3.207 to 8.593]
Statistical Analysis 2: Comparison: Bimekizumab 320 mg Q4W + Bimekizumab 320 mg Q4W/Q8W (RS) vs Adalimumab (RS); [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-values for the comparison of treatment groups were based on the CMH test from the general association; Odds Ratio (OR) = 4.974, 95% CI 2-sided [3.257 to 7.594]

8. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 56
Description: PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline. Body divided into 4 areas: head/arms/trunk to groin/and legs to top of buttocks. Assignment of an average score for the redness/thickness/scaling for each of the 4 body areas with a score of 0 (clear)-4 (very marked). Determining the percentage of skin covered with PSO for each of the body areas and converting to a 0-6 scale. Final PASI=average redness/thickness/scaliness of the psoriatic skin lesions multiplied by the involved psoriasis area score of the respective section and weighted by the percentage of the person's affected skin for the respective section. The min possible PASI score is 0=no disease, max score is 72=maximal disease.
Time Frame: Week 56
Population: The RS consisted of all randomized study participants. ADA participants were not included as they did not start BKZ treatment at Baseline, thus did not have a year of BKZ treatment. The purpose of this table is to look at response after one year of BKZ.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W/Q8W (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 161 | 158
percentage of participants | 82.6 | 84.8

9. Secondary Outcome: Percentage of Participants With an IGA Response (Clear or Almost Clear With at Least 2-category Improvement Relative to Baseline) at Week 56
Description: IGA measures the overall psoriasis severity following a 5-point scale (0-4), where scale 0=clear, no signs of psoriasis; presence of post-inflammatory hyperpigmentation, scale 1=almost clear, no thickening; normal to pink coloration; no to minimal focal scaling, scale 2=mild thickening, pink to light red coloration and predominately fine scaling, 3=moderate, clearly distinguishable to moderate thickening; dull to bright red, clearly distinguishable to moderate thickening; moderate scaling and 4=severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions. IGA response was defined as clear [0]/almost clear [1] with at least a 2-category improvement from Baseline at Wk56.
Time Frame: Week 56
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 320 mg Q4W/Q8W (RS) | Bimekizumab 320 mg Q4W (RS)
Number analyzed (Participants) | 161 | 158
percentage of participants | 83.2 | 82.3

10. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Week 24
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to Week 24
Population: The Safety Set (SS) consisted of all study participants who received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS): Participants received bimekizumab 320 mg Q4W for 16 weeks and proceeded with bimekizumab 320 mg Q8W until Week 24. Participants received placebo at pre-specified time-points to maintain the blinding. Participants formed the Safety Set (SS).
- Bimekizumab 320 mg Q4W Through Week 24 (SS): Participants received bimekizumab 320 mg Q4W for 24 weeks. Participants received placebo at pre-specified time-points to maintain the blinding. Participants formed the SS.
- Adalimumab Through Week 24 (SS): Participants received adalimumab for 24 weeks. Participants received placebo at pre-specified time-points to maintain the blinding. Participants formed the SS.
Arm/Group | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) | Bimekizumab 320 mg Q4W Through Week 24 (SS) | Adalimumab Through Week 24 (SS)
Number analyzed (Participants) | 161 | 158 | 159
no. of new events per 100 subject-years | 310.44 [256.52 to 372.34] | 300.71 [247.60 to 361.83] | 297.54 [244.77 to 358.31]

11. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Week 24
Description: The number of SAEs adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to Week 24
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) | Bimekizumab 320 mg Q4W Through Week 24 (SS) | Adalimumab Through Week 24 (SS)
Number analyzed (Participants) | 161 | 158 | 159
no. of new events per 100 subject-years | 1.37 [0.03 to 7.66] | 5.61 [1.53 to 14.38] | 6.98 [2.27 to 16.30]

12. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Week 24
Description: The number of TEAEs leading to discontinuation adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to Week 24
Population: The Safety Set (SS) consisted of all study participants that received at least 1 dose of IMP.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) | Bimekizumab 320 mg Q4W Through Week 24 (SS) | Adalimumab Through Week 24 (SS)
Number analyzed (Participants) | 161 | 158 | 159
no. of new events per 100 subject-years | 8.30 [3.05 to 18.07] | 4.16 [0.86 to 12.17] | 6.98 [2.27 to 16.29]

13. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Safety Follow-Up Visit (up to Week 72)
Description: The number of TEAEs adjusted by duration of exposure to study treatment was scaled such that it provided an incidence rate per 100 patient-years. If a participant had multiple events, the time of exposure was calculated to the first occurrence of the AE being considered. If a participant had no events, the total time at risk was used.
Time Frame: From Baseline to Safety Follow-Up Visit (up to Week 72)
Population: The Bimekizumab Set (BKZ Set) consisted of all study participants who received at least 1 dose of bimekizumab in this study.
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Groups:
- Any Bimekizumab 320 mg Q8W (BKZ Set): This arm consisted of all participants who received bimekizumab 320 mg Q8W at any time in the study (up to 56 weeks). Participants formed the bimekizumab Set (BKZ Set).
- Any Bimekizumab 320 mg Q4W (BKZ Set): This arm consisted of all participants who received bimekizumab 320 mg Q4W at any time in the study (up to 56 weeks). Participants formed the bimekizumab Set (BKZ Set).
Arm/Group | Any Bimekizumab 320 mg Q8W (BKZ Set) | Any Bimekizumab 320 mg Q4W (BKZ Set)
Number analyzed (Participants) | 154 | 468
no. of new events per 100 subject-years | 231.38 [191.68 to 276.88] | 262.41 [235.37 to 291.71]

14. Secondary Outcome: Number of Serious Adverse Events (SAEs) Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Safety Follow-Up Visit (up to Week 72)
Description: as for outcome 11
Time Frame: From Baseline to Safety Follow-Up Visit (up to Week 72)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Any Bimekizumab 320 mg Q8W (BKZ Set) | Any Bimekizumab 320 mg Q4W (BKZ Set)
Number analyzed (Participants) | 154 | 468
no. of new events per 100 subject-years | 7.03 [3.04 to 13.86] | 5.34 [3.05 to 8.67]

15. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal Adjusted by Duration of Participant Exposure to Study Treatment From Baseline to Safety Follow-Up Visit (up to Week 72)
Description: as for outcome 12
Time Frame: From Baseline to Safety Follow-Up Visit (up to Week 72)
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: no. of new events per 100 subject-years
Arm/Group | Any Bimekizumab 320 mg Q8W (BKZ Set) | Any Bimekizumab 320 mg Q4W (BKZ Set)
Number analyzed (Participants) | 154 | 468
no. of new events per 100 subject-years | 4.37 [1.42 to 10.19] | 4.62 [2.53 to 7.75]

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were collected from Baseline to Safety Follow-Up Visit (up to Week 72)
Description: Treatment-emergent AEs were defined as those AEs that had a start date on or following the first dose of study treatment through the final dose of study treatment + 140 days (covering up to Safety Follow-Up Visit for study participants not enrolling in Open-label Extension (OLE) study).
Arm/Group | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) | Bimekizumab 320 mg Q4W Through Week 24 (SS) | Adalimumab Through Week 24 (SS) | Any Bimekizumab 320 mg Q8W (BKZ Set) | Any Bimekizumab 320 mg Q4W (BKZ Set)
All-Cause Mortality (participants affected / at risk) | 0/161 | 0/158 | 1/159 | 0/154 | 0/468
Serious Adverse Events (participants affected / at risk) | 1/161 | 4/158 | 5/159 | 8/154 | 16/468
Other Adverse Events (participants affected / at risk) | 65/161 | 61/158 | 62/159 | 60/154 | 182/468
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) (N=161) | Bimekizumab 320 mg Q4W Through Week 24 (SS) (N=158) | Adalimumab Through Week 24 (SS) (N=159) | Any Bimekizumab 320 mg Q8W (BKZ Set) (N=154) | Any Bimekizumab 320 mg Q4W (BKZ Set) (N=468)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Infected dermal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Helicobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 320 mg Q4W/Q8W Through Week 24 (SS) (N=161) | Bimekizumab 320 mg Q4W Through Week 24 (SS) (N=158) | Adalimumab Through Week 24 (SS) (N=159) | Any Bimekizumab 320 mg Q8W (BKZ Set) (N=154) | Any Bimekizumab 320 mg Q4W (BKZ Set) (N=468)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 8 (9) | 4 (6) | 5 (5) | 14 (16)
Nasopharyngitis (Infections and infestations) | 27 (40) | 32 (46) | 38 (50) | 28 (35) | 79 (113)
Oral candidiasis (Infections and infestations) | 19 (26) | 15 (20) | 0 (0) | 17 (26) | 66 (104)
Upper respiratory tract infection (Infections and infestations) | 12 (14) | 7 (8) | 15 (21) | 13 (16) | 30 (40)
Pharyngitis (Infections and infestations) | 5 (7) | 4 (4) | 1 (1) | 11 (11) | 13 (14)
Hypertension (Vascular disorders) | 9 (10) | 6 (6) | 13 (13) | 4 (4) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/47/NCT03412747/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT03412747/SAP_001.pdf